CLINICAL TRIAL: NCT05563389
Title: the Impact of Statin on Cirrhotic Patients
Brief Title: Statin Impact on Hepatic Decompensation
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Khadija Ahmed Mhrose Glal, Assistant lecturer of clinical pharmacy- Clinical pharmacy department- Faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Statin and iver cirrhosis
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Quality of Life
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLACEBO (Placebo Comparator): placebo formula
  Interventions: Drug: Placebo
- statin (Active Comparator): atorvastatin tablets
  Interventions: Drug: Atorvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 20mg — active arm
  Other Names: atorvastatin
  Arms: statin
Drug: Placebo — placebo arm
  Arms: PLACEBO

SUMMARY:
The study aims to evaluate the impact of statin on hepatic decompensation.

DETAILED DESCRIPTION:
Cirrhosis is the late stage of liver damage and possess two phases:. The shift from compensated to decompensated cirrhosis is characterized by the onset of complications) which are associated with substantial morbidity and negative Impact on quality of life (QOL)Cirrhosis and its complications have a substantial economic, social, and personal impact on affected patients, as well as their families and caregivers

ELIGIBILITY:
Inclusion Criteria:

* cirrhosis adult both sex

Exclusion Criteria:

* renal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

PRIMARY OUTCOMES:
impact on decompensation | 6 months
  change in recurrence of cirrhosis related complications

CONTACTS AND LOCATIONS:
Overall Officials: khadija glal, Principal Investigator — assistant lecturer
Locations (1):
- Tanta University, Tanta, Egypt